CLINICAL TRIAL: NCT02981719
Title: Simultaneous Gemcitabine and Irreversible Electroporation for Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y2016-MS-001
Record Dates: First submitted 2016-10-31; First posted 2016-12-05 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simultaneous gemcitabine and irreversible electroporation (Experimental): gemcitabine intravenous infusion prior to irreversible electroporation treatment.
  Interventions: Procedure: simultaneous gemcitabine and irreversible electroporation
- IRE group (Other): percutaneous irreversible electroporation for locally advanced pancreatic cancer.
  Interventions: Procedure: irreversible electroporation

INTERVENTIONS:
Procedure: simultaneous gemcitabine and irreversible electroporation — gemcitabine intravenous infusion prior to irreversible electroporation treatment
  Arms: simultaneous gemcitabine and irreversible electroporation
Procedure: irreversible electroporation — percutaneous irreversible electroporation was performmed for locally advaanced pancreatic cancer.
  Arms: IRE group

SUMMARY:
The aim of this study was to compare the therapeutic efficacy between simultaneous gemcitabine administration and IRE and IRE alone for locally advanced pancreatic cancer (LAPC)

DETAILED DESCRIPTION:
in the GEM- IRE group, before the IRE ablation started, patients received 1000 mg/m2 gemcitabine hydrochloride [Qilu pharmaceutical (Hainan) Co., Ltd. Haikou, China] intravenously (over approximately 30 min).

In the IRE group, the IRE ablation was performed without gemcitabine intravenous infusion before IRE.

The aim of this study was to evslusted the overall survival (OS), objective response rate (ORR) and adverse events after simultaneous therapy.

ELIGIBILITY:
Inclusion Criteria:

* Radiologic confirmation of unresectable locally advanced pancreatic cancer by at least CT of chest and abdomen
* Screening must be performed no longer than 2 weeks prior to study inclusion
* Maximum tumor diameter ≤ 5 cm
* Histological or cytological confirmation of pancreatic adenocarcinoma;
* Age ≥ 18 years
* PS-classification 0 - 2
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to definite inclusion;
* Hemoglobin level ≥ 115 g/L
* Platelet count ≥ 100*109/l
* Neutrophil count ≥ 2×109/L;
* White blood cell count ≥ 4 ×109/L;
* ALT and AST ≤ 2.5 x ULN
* Serum creatinine ≤ 1.5 x ULN or a calculated creatinine clearance ≥ 50 ml/min
* Prothrombin time or INR < 1.5 x ULN
* Written informed consent

Exclusion Criteria:

* Resectable pancreatic adenocarcinoma as discussed by our multidisciplinary hepatobiliary team
* History of epilepsy
* History of cardiac disease:
* Cardiac arrhythmias requiring anti-arrhythmic therapy or pacemaker (beta blockers for antihypertensive regimen are permitted)
* Compromised liver function (e.g. signs of portal hypertension, INR > 1,5 without use of anticoagulants, ascites)
* Uncontrolled infections (> grade 2 NCI-CTC version 3.0)
* Pregnant. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment
* Allergy to contrast media
* Any implanted stimulation device
* Any implanted metal stent/device within the area of ablation that cannot be removed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Safety (number of adverse effects) | 3 month
  Adverse events

SECONDARY OUTCOMES:
Tumor response | 12 months
  Imaging evaluation
Overall survival (OS) | 36 months
  Overall survival (OS) was defined using time of death.
Carbohydrate antigen 19-9 (CA19-9) | 1 month
  carbohydrate antigen 19-9 (CA19-9) levels were measured.
Technical success of ablation | 3 months
  The technical success addressed whether the tumor was treated according to protocol and was covered completely by the ablation zone.

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, PHD, Study Chair — Fuda Cancer Hospital
Locations (1):
- FUDA Cancer Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided